CLINICAL TRIAL: NCT01463566
Title: Prospective Multicenter Post-market Study of the Zimmer Gender Solutions Natural Knee Flex System
Brief Title: Gender Solutions Natural Knee Post-Market Study
Status: Withdrawn | Type: Observational
Why Stopped: Suspended pending internal review/direction of the company's focus.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CMU2011-05K
Record Dates: First submitted 2011-10-24; First posted 2011-11-02 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis; Inflammatory Arthritis; Post-traumatic Arthritis; Rheumatoid Arthritis; Osteonecrosis; Varus or Valgus Deformities
Keywords: arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis; Arthritis, Rheumatoid; Osteonecrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 - Gender Natural Knee: Patients suffering from severe knee pain and disability.
  Interventions: Device: Zimmer Gender(R) Solutions(TM) Natural-Knee(R) Flex System

INTERVENTIONS:
Device: Zimmer Gender(R) Solutions(TM) Natural-Knee(R) Flex System — Gender Solutions Natural Knee Flex System in total knee arthroplasty

SUMMARY:
This is a prospective multicenter study of the Gender Solutions Natural Knee Flex System when used in primary total knee arthroplasty. The purpose of the study is to obtain short-, Mid-, and long-term clinical outcomes and implant survivorship data for the Gender Solutions Natural Knee Flex System.

DETAILED DESCRIPTION:
Survival and outcome data on the Gender Solutions Natural Knee Flex System will be done by an analysis of standard scoring system, radiographs and adverse event records. Survivorship will be evaluated by monitoring the frequency and incidence of adverse events, serious adverse events, adverse device effects, serious adverse device effects, and unanticipated adverse device effects. Outcomes will be measured by comparing the overall pain and function performances (based on the Knee Society Scoring System), survivorship, subject quality of life and radiographic parameters of study subjects receiving the Gender Solutions Natural Knee Flex System.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18-75 years of age, inclusive;
* Patient qualifies for a total knee arthroplasty based on physical exam and medical history including at least one of the following: osteoarthritis, inflammatory arthritis, post-traumatic arthritis, rheumatoid arthritis, or valgus, varus, or flexion deformities;
* Patient has undergone a study related informed consent process;
* Patient is willing and able to provide written consent;
* Patient is willing and able to cooperate in the required post-operative therapy;
* Patient is willing and able to complete scheduled follow-up evaluations.

Exclusion Criteria:

* Patient has previous history of infection in the affected joint and/or a local or systemic infection that could affect the prosthetic joint;
* Insufficient bone stock on femoral or tibial surfaces;
* Skeletal immaturity
* Neuropathic arthropathy
* Osteoporosis or any loss of musculature or neuromuscular disease that compromises the affected limb;
* Stable, painless arthrodesis in a satisfactory functional position;
* Severe instability secondary to the absence of collateral ligament integrity;
* Patient has rheumatoid arthritis and an ulcer of the skin or a history of recurrent breakdown of the skin because of their risk of postoperative infection is greater;
* Patient has known sensitivity or allergy to one or more of the implanted materials;
* Patients pregnant or considered a member of a protected population (e.g., prisoner, mental incompetence, unable to understand what clinical trial participation entails, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each investigator will screen from his patient population patients suffering from severe knee pain and disability who meet the inclusion/exclusion criteria for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2024-07 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Survivorship | 10 years
  Based on frequency of adverse events, serious adverse events, adverse device effects, serious adverse devices effects and unanticipated adverse device effects or removal of the device summarized using a Kaplan-Meier method and presented with rates (as percentages) and confidence intervals.

SECONDARY OUTCOMES:
Pain Performance | 10 years
  Measured by comparing the overall pain performances (based on Knee Society Scoring System), Survivorship, subject quality of life and radiographic parameters.
Function Performance | 10 Years
  Measured by comparing the overall function performances (based on the Knee Society Scoring System), survivorship, subject quality of life and radiographic parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Kacy Arnold, RN, MBA, Study Director — Zimmer Biomet